CLINICAL TRIAL: NCT00403403
Title: A Placebo-Controlled, Double-Blind, Multicenter, Randomized, Phase II Study of Bevacizumab in Previously Untreated Extensive-Stage Small Cell Lung Cancer
Brief Title: A Study of Bevacizumab in Previously Untreated Extensive-Stage Small Cell Lung Cancer (SALUTE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: David Karlin, M.D., Study Director, Genentech, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVF3995g
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Results first posted 2011-02-25 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Small Cell Lung Cancer
Keywords: SCLC; SALUTE; Lung Cancer; Avastin
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms | interventions — Bevacizumab; Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo+Chemotherapy (Placebo Comparator): Chemotherapy = cisplatin (or carboplatin) + etoposide
  Interventions: Drug: Chemotherapy; Drug: Placebo
- Bevacizumab+Chemotherapy (Experimental): Chemotherapy = cisplatin (or carboplatin) + etoposide
  Interventions: Drug: Bevacizumab; Drug: Chemotherapy

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab 15 mg/kg by intravenous (IV) infusion on Day 1 of each of the first four 21-day cycles during chemotherapy, followed by single agent administration until disease progression, unacceptable toxicity, discontinuation from study, or death.
  Arms: Bevacizumab+Chemotherapy
Drug: Chemotherapy — Chemotherapy = cisplatin (or carboplatin) + etoposide. Cisplatin 75 mg/m² IV on Day 1 of each of the first four 21-day cycles OR carboplatin (area under the curve [AUC]=5 mg/mL/min, per Calvert formula) IV on Day 1 of each of the first four 21-day cycles; etoposide 100 mg/m² on Days 1-3 of each of the first four 21-day cycles.
Drug: Placebo — Placebo 15 mg/kg by intravenous (IV) infusion on Day 1 of each of the first four 21-day cycles during chemotherapy, followed by single agent administration until disease progression, unacceptable toxicity, discontinuation from study, or death.
  Arms: Placebo+Chemotherapy

SUMMARY:
This is a placebo-controlled, double-blind, multicenter, randomized study for preliminary evaluation of the efficacy and safety of combining bevacizumab with cisplatin (or carboplatin) and etoposide in patients with previously untreated extensive-stage small cell lung cancer (SCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented small cell carcinoma of the bronchus, classified as extensive-stage disease
* Measurable disease or lesions
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2

Exclusion Criteria:

* Life expectancy of < 12 weeks
* Current, recent, or planned participation in another experimental drug study
* Ongoing or active infection
* Active malignancy other than SCLC or superficial basal/squamous cell carcinoma within the previous 5 years
* Prior systemic therapy, radiation therapy, or surgery for SCLC
* Inadequate bone marrow function, renal function, or hepatic function
* Serum sodium of < 120 mg/dL
* Inadequately controlled hypertension
* History of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association Class II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to study enrollment
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* Known central nervous system disease, except for brain metastases treated with whole-brain radiotherapy
* Significant vascular disease or recent peripheral arterial thrombosis within 6 months prior to study enrollment
* History of hemoptysis within 4 weeks prior to study enrollment
* Evidence of bleeding diathesis or coagulopathy in the absence of therapeutic anticoagulation
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of a need for a major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, including placement of a vascular access device, within 7 days prior to Day 1
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to study enrollment
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Known hypersensitivity to any component of bevacizumab
* Pregnant (positive pregnancy test) or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2007-03; Primary Completion 2009-02 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Karlin, M.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo+Chemotherapy: Chemotherapy = cisplatin (or carboplatin) + etoposide. Placebo 15 mg/kg by intravenous (IV) infusion on Day 1 of each of the first four 21-day cycles during chemotherapy, followed by single agent administration until disease progression, unacceptable toxicity, discontinuation from study, or death. Cisplatin 75 mg/m² IV on Day 1 of each of the first four 21-day cycles OR carboplatin (area under the curve [AUC]=5 mg/mL/min, per Calvert formula) IV on Day 1 of each of the first four 21-day cycles; etoposide 100 mg/m² on Days 1-3 of each of the first four 21-day cycles.
- Bevacizumab+Chemotherapy: Chemotherapy = cisplatin (or carboplatin) + etoposide. Bevacizumab 15 mg/kg by intravenous (IV) infusion on Day 1 of each of the first four 21-day cycles during chemotherapy, followed by single agent administration until disease progression, unacceptable toxicity, discontinuation from study, or death. Cisplatin 75 mg/m² IV on Day 1 of each of the first four 21-day cycles OR carboplatin (area under the curve [AUC]=5 mg/mL/min, per Calvert formula) IV on Day 1 of each of the first four 21-day cycles; etoposide 100 mg/m² on Days 1-3 of each of the first four 21-day cycles.
Period: Overall Study
Arm/Group | Placebo+Chemotherapy | Bevacizumab+Chemotherapy
Started | 50 | 52
Safety-Evaluable Patients | 47 | 51
Completed | 50 | 52
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo+Chemotherapy | Bevacizumab+Chemotherapy | Total
Number analyzed (Participants) | 50 | 52 | 102
Age Continuous [Mean (Standard Deviation); unit: years] | 64.0 (10.0) | 61.3 (8.5) | 62.7 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 26 | 46
  Male | 30 | 26 | 56

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Duration of PFS, defined as the time from randomization to disease progression or on-study death, whichever occurred first.
Time Frame: Randomization until progression or lost to follow-up (up to 2 years)
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo+Chemotherapy | Bevacizumab+Chemotherapy
Number analyzed (Participants) | 50 | 52
Months | 4.4 [4.2 to 4.9] | 5.5 [4.5 to 6.7]
Statistical Analysis 1: Comparison: Placebo+Chemotherapy vs Bevacizumab+Chemotherapy; Test type: Superiority or Other; p = 0.0097, Log Rank; Hazard Ratio (HR) = 0.528, 95% CI [0.323 to 0.862] — HR estimated from a stratified Cox regression model, stratified for ECOG performance (0-1 vs. 2) and chemotherapy type (cisplatin vs. carboplatin)

2. Secondary Outcome: Overall Survival
Description: Duration of overall survival from randomization until death or loss to follow-up
Time Frame: Randomization until death or lost of follow-up (up to 27 months)
Population: Intent-to-treat population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo+Chemotherapy | Bevacizumab+Chemotherapy
Number analyzed (Participants) | 50 | 52
Months | 10.9 [8.1 to 14.7] | 9.4 [8.7 to 11.3]
Statistical Analysis 1: Comparison: Placebo+Chemotherapy vs Bevacizumab+Chemotherapy; Test type: Superiority or Other; p = 0.6054, Log Rank; Hazard Ratio (HR) = 1.160, 95% CI 2-sided [0.660 to 2.039] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants With an Objective Response
Description: Objective response was defined as a complete or partial response (per RECIST) determined by two investigator assessments conducted at least 4 weeks apart.
  Complete Response (CR), Partial Response (PR), Incomplete Response (IR), Stable Disease (SD) (per RECIST):
  Target Lesions Non-Target Lesions New Lesions Overall Response CR CR No CR CR IR/SD No PR PR Non-PD No PR
Time Frame: Randomization until progression or lost to follow-up (up to 2 years)
Population: Intent-to-treat population
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo+Chemotherapy | Bevacizumab+Chemotherapy
Number analyzed (Participants) | 50 | 52
Percentage of participants | 48.0 | 57.7
Statistical Analysis 1: Comparison: Placebo+Chemotherapy vs Bevacizumab+Chemotherapy; Test type: Superiority or Other; p = 0.3269, Chi-squared; Mean Difference (Final Values) = 9.7, 95% CI [-9.6 to 29.0]

4. Secondary Outcome: Number of Participants With an Objective Response
Description: as for outcome 3
Time Frame: Randomization until progression or lost to follow-up (up to 2 years)
Measure: Number; unit: number of participants
Arm/Group | Placebo+Chemotherapy | Bevacizumab+Chemotherapy
Number analyzed (Participants) | 50 | 52
number of participants | 24 | 30

5. Secondary Outcome: Duration of Objective Response
Description: Duration of response was defined as time from the first response date to disease progression or on-study death (i.e., death occurring any time from randomization to 30 days after the final treatment with bevacizumab/placebo). Objective response was defined as a complete or partial response (per RECIST) determined by two investigator assessments conducted at least 4 weeks apart.
Time Frame: Randomization until progression or lost to follow-up (up to 2 years)
Population: Randomized patients with measurable disease at baseline.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Placebo+Chemotherapy | Bevacizumab+Chemotherapy
Number analyzed (Participants) | 24 | 30
Months | 3.2 [2.9 to 4.2] | 4.7 [4.2 to 5.8]
Statistical Analysis 1: Comparison: Placebo+Chemotherapy vs Bevacizumab+Chemotherapy; Test type: Superiority or Other; p = 0.0011, Log Rank; Hazard Ratio (HR) = 0.305, 95% CI 2-sided [0.144 to 0.644] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Overall duration of study
Description: Safety analyses were performed on the safety evaluable population, which included 98 patients who received at least one dose of chemotherapy, bevacizumab, or placebo.
  National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)
Arm/Group | Placebo+Chemotherapy | Bevacizumab+Chemotherapy
Serious Adverse Events (participants affected / at risk) | 11/47 | 20/51
Other Adverse Events (participants affected / at risk) | 31/47 | 35/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo+Chemotherapy (N=47) | Bevacizumab+Chemotherapy (N=51)
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0
Pericardial Effusion (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 2
Gastrointestinal Perforation (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 3
Lobar Pneumonia (Infections and infestations) | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0
Hemoglobin Decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Depressed Level of Consciousness (Nervous system disorders) | 0 | 1
Reversible Posterior Leukoencephalopathy Syndrome (Nervous system disorders) | 0 | 1
Mental Status Changes (Psychiatric disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo+Chemotherapy (N=47) | Bevacizumab+Chemotherapy (N=51)
Neutropenia (Blood and lymphatic system disorders) | 20 | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 4
Hypertension (Vascular disorders) | 12 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.